CLINICAL TRIAL: NCT02264366
Title: ACCELERATION: An Activity,Smoking Cessation, Healthy Eating and Alcohol Intervention Program With Motivational Supports Aimed at Chronic Disease Prevention
Brief Title: Activity ,Smoking Cessation, Healthy Eating and Alcohol Intervention Program:(ACCELERATION)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Nova Scotia Health Authority (Other); Sunnybrook Health Sciences Centre (Other); University of British Columbia (Other); Concordia University, Montreal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACCELERATION
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- At Risk Group: ACCELERATION program (Experimental): This "At Risk" Group will include ;People at risk of cancer referred from UHN partners and community practices. Also included in this group are; First Nations population of BC, Asians and South Asian populations from Greater Vancouver and the working population of the City of Richmond employees. At the Montreal site users of the YMCA with risk factors for, or family history of, cancer and other chronic diseases will be targeted. And finally, in Nova Scotia the "At Risk" Group will be identified as being at risk of cancer and other chronic diseases referred from community practices and from the workplace population of the Capital District Health Authority (CDHA).
  Intervention: Motivational Communication for Health Behavior management
  Interventions: Behavioral: Motivational Communication for Health Behavior management
- Friends & Family -ACCELERATION Program (Experimental): This group includes family and friends of cancer survivors and family and friends of cardiac & COPD rehab patients. The intervention includes Motivational Communication for Health Behavior management
  Interventions: Behavioral: Motivational Communication for Health Behavior management

INTERVENTIONS:
Behavioral: Motivational Communication for Health Behavior management — An appropriate and evidence-informed model of motivational counselling, health coaching and chronic disease self-management will be integrated into the delivery of all aspects of the ACCELERATION program. The focus will be on 4 health behaviors that include healthy eating, exercise, smoking cessation and moderation of alcohol consumption. This will include engagement techniques such as motivational interviewing, identification of stage of change, visioning of "best self", goal setting and action planning, expressing empathy, developing discrepancy, decisional balance, "rolling with resistance", and supporting self-efficacy. (Rubak 2005, Knight 2006).
  Other Names: Behavior Change

SUMMARY:
The ACCELERATION (ACtivity, smoking Cessation, healthy Eating and aLcohol Education, inteRvention, and motivATION) Program is a collaborative project in cancer and chronic disease prevention that has been designed by and will be delivered amongst cardiopulmonary rehabilitation and prevention programs and cancer centres in Ontario (ON), British Columbia (BC), Quebec (QC) and Nova Scotia (NS). This project is being funded by the Canadian Partnership Against Cancer, Health Canada and Heart and Stroke Foundation of Canada and in the amount of $2.4M over a 3 year period (October 2013 - September 2016). The ACCELERATION Program is a 12 week structured model of behavioural interventions and education around self-management and prevention that aims to access readily available and referable people for primary prevention intervention.This program aligns with current provincial, national and international chronic disease prevention and management strategies. The goal of the ACCELERATION program is to measurably and effectively change the risk factors and health behaviours known to impact cancer and other chronic diseases. Specifically we will aim to increase physical activity, reduce smoking, encourage healthy eating, and moderate alcohol consumption in about 3,000 participants across Canada over 3 years.

DETAILED DESCRIPTION:
Chronic diseases including cancer, cardiovascular disease, lung conditions and diabetes are the leading cause of mortality and morbidity in Canada and worldwide. These chronic conditions share common modifiable risk factors including physical inactivity, suboptimal nutrition, smoking and excessive alcohol intake. Cardiac rehabilitation centres in this Coalition have been providing primary and secondary prevention services for many years focused on these behavioural risks, and many of our participants with heart disease also have co-morbidities including cancer, diabetes and lung disease. Co-morbidities are a clinical reality, and we no longer deal with diseases singularly. Today, our client population is more diverse than ever and fiscal constraints call for the pooling of prevention resources to simultaneously address a range of chronic diseases impacted by common risk factors.

Extending our reach to populations at risk of cancer and other chronic diseases, populations which are readily available and referable In Ontario, UHN/Toronto Rehab has a cancer program for women who have survived breast cancer as well as women undergoing cancer treatment. Discussions with Princess Margaret Hospital point to opportunities to extend programming to more cancer patients and people at risk of cancer. The ELLICSR arm of Princess Margaret Hospital, which focuses on helping survivors, has expressed interest in collaborating to reach family and friends of cancer survivors, for primary prevention. Likewise, the Odette Cancer Centre at Sunnybrook Hospital sees over 900 new women every year who are referred due to a family history of breast cancer. They have expressed to us that they can identify and will refer women at high risk of developing breast cancer into our proposed primary prevention program. Similarly, in Quebec, L'Hôpital du Sacré-Cœur de Montréal has one of the nation's highest rated lung cancer groups. Our Quebec partner, Centre de réadaptation cardio-respiratoire Jean-Jacques-Gauthier (CRJJG) has strong ties to this program. With funding, they will be able to reach and deliver prevention programmes to the family and friends of their lung cancer clients, an opportunity that exists because family and friends tend to be more engaged and open to the possibility of lifestyle change.

This is why we have partnered with these cancer centres in this Coalition: to formalize our existing partnerships and focus our resources on the population at risk of cancer that is readily available and referable for primary prevention.

The links that our Coalition partners have with primary care hold opportunities not yet seized. In Ontario, the Department of Family and Community Medicine at Sunnybrook has many patients at risk for, or with, multiple chronic diseases.

The opportunity that exists to reach pregnant women with obesity-related risks is one that could be seized Canada-wide. The unfortunate reality is that obesity complicates about 50% of pregnancies today.

The opportunity, and need, to impact a person's family and social circle Our program concept is founded on the idea that 'you really need to get the whole family' to sustain the long-term impact of prevention and change in behaviour. We know there is evidence that family/social support can help. A systematic review on childhood obesity identified promising strategies that included parent support and home activities that encourage children to be more active, eat more nutritious foods and spend less time in screen-based activities (Waters et al, 2011).

As Lead Agency, the UHN/Toronto Rehab already runs a successful Cardiac Rehab @ Home program which is a six-month program that sees approximately 120 clients per year. The average client lives approximately 200kms away from the urban area, is younger, and more likely to be working, compared to on-site clients. An evaluation has shown that the program is effective with similar outcomes as an on-site program: clients made the same gains in cardiovascular fitness and were just as likely to adhere to the program. The study also showed that such programs are more cost-effective than on-site programs for participants living in remote areas (Scane et al, 2012).

Deepening and broadening our reach to selected at risk populations already connected to us.

Many of the core partners not only have links to their local communities but have years of collaboration with the community on prevention. Notably, our BC partner, the BC Cardiovascular Physiology & Rehabilitation Laboratory, has extensive primary prevention experience having worked with more than 300,000 participants in the past 10 years on community-based programs for children (school-based and out-of-school), workplace wellness (e.g. police and firefighters) and population groups at risk for chronic disease.

Additionally, they have solid partnerships with Aboriginal communities throughout BC. Formal partnerships have been forged with Aboriginal communities throughout BC including extensive research in rural and remote communities.

Through the Coalition's work and history with the Aboriginal communities, and because they know there is evidence that there are health benefits for Aboriginal peoples in participating in a community-based physical activity intervention , the ACCELERATION program could be delivered with relative ease to these communities in BC.

The Centre de réadaptation cardio-respiratoire Jean-Jacques-Gauthier (CRJJG) provides prevention programming for patients with cardiovascular (heart disease and heart failure) and respiratory disease (chronic obstructive pulmonary disease and asthma). One very unique aspect is the ongoing asthma prevention work of this coalition member. This adult asthma population are, on average, younger than most classical rehabilitation groups (ca. 40 years old) and, whilst not having overt cancer or cardiovascular disease, do normally display several risk factors, which provides a model of engaging and adapting the ACCELERATION program to these kinds of populations.

Furthermore, the CRJJG is conveniently housed within the YMCA Cartierville. There is, therefore, already a strong partnership with the YMCA. The proposed program will allow our Quebec partner to deliver a prevention program to YMCA users with risk factors or a family history of chronic diseases. In addition, the YMCA Cartierville has a unique partnership with the local council where it provides free access to non-YMCA local community members, thus allowing the ACCELERATION programme to be delivered to a very diverse cultural and socio-economic community base.

Finally, the CRJJG has specific expertise in motivational interviewing (MI) , which is a client-centred communication tool focusing on enhancing intrinsic motivation to change a particular behaviour, and exploring and resolving ambivalence about behavior change (Lavoie et al, 2012).

At the Eastern end of Canada, the province of Nova Scotia has one of the highest rates of cardiovascular disease in the country with a prevalence of 6.4% (Heart and Stroke Foundation, 2012). There is also an excess incidence and prevalence of lung, colorectal, prostate, melanoma and breast cancer (Canadian Cancer Society). This is one reason we chose to partner with Nova Scotia. Our partner runs the Community Cardiovascular Hearts in Motion (CCHIM) program which is a community-based exercise and health education program. Referrals are accepted from predominantly family doctors but also other specialists and allied health professionals including physiotherapists, nurse practitioners and diabetes clinics. Patients expand the complete vascular spectrum from primary care to all levels of secondary prevention. There is also a Heart Health Clinic available to assist those individuals living with more complicated and higher risk cardiac and pulmonary disease (tertiary). The successes of this program are translatable to the ACCELERATION program that targets people at risk of cancer and chronic diseases, as well as family and friends of people who have suffered an acute event associated with a chronic disease.

Our Nova Scotia partner notes that there is strong representation of females in the primary prevention arm of CCHIM and most of these are obese with diabetes. The planned Ontario program with ante- and post-partum women at risk of obesity-related cancer is replicable for the Nova Scotia female population, and we would seek to transfer knowledge and replicate the program in Nova Scotia as well.

There is also an opportunity to reach the underserviced black population. Incidence rate ratios for African Canadians relative to the general population of Nova Scotia were significantly elevated for circulatory disease, diabetes and psychiatric disorders (Kisely et al, 2008). Our Nova Scotia partner (CCHIM) sees opportunity in providing a virtual program for this population. CCHIM is in present development of translational research to move beyond the "bricks and mortar" to reach such patient populations who are in need of such a program by virtue of risk or established disease but cannot, or will not, attend. This will be run through the primary care physician and local health care teams (such as NP clinics, addiction services, etc). It will allow for adaptation and implementation when the patient is "ready" to engage (similar to smoking cessation as per the "Ottawa Model"). This approach will be adapted to the present project in an effort to expand its exposure further while evaluating the elements that are sustainable upon project completion.

In Ontario, the South Asian population is the largest visible minority group in Ontario, and one with a higher prevalence of chronic diseases compared to other groups (Statistics Canada, 2010; Fraser Health, 2013). They would benefit from a targeted program like ACCELERATION that is customized for them, and made culturally appropriate to their beliefs, values and customs.

Deepening prevention impact in workplaces Two of our key partners (BC and NS) have existing partnerships with large employers.

In BC, our partner has a formal research relationship with the City of Richmond. They evaluate the risk for chronic disease in approximately 200-300 City of Richmond workers each year. The proposed program will allow the introduction of a workplace wellness program for these workers. We estimate that with the awarding of this program that the current workplace wellness program will expand meeting the needs of family and friends of city workers meeting a direct mandate of the City of Richmond employers.

Our Nova Scotia partner will engage their Capital District Health Authority (CDHA) workplace, drawing participants from a population of 10,000 employees. Having both a set program and a virtualization of the program will offer a unique opportunity to address both the benefits to at risk patients as well as the application of a program to the most common yet possibly the most difficult workplace sector to access.

ELIGIBILITY:
Inclusion Criteria:

Must have at least one behavioural risk factor

* physical inactivity (less than 150 minutes of moderate to vigorous physical activity per week)
* suboptimal nutrition behaviour (consumption of less than 5 fruits/vegetables per day)
* smoking (any amount of personal smoking by self-report)
* alcohol intake in excess of Canada's Low-Risk Alcohol Drinking Guidelines (low risk is defined by less than 10 drinks a week for women, with no more than 2 drinks a day most days; or less than 15 drinks a week for men, with no more than 3 drinks a day most days)
* over the age of 18
* family history of cancer or cardiovascular disease
* in addition, subjects may have stable medical co-morbidities such as hypertension, dyslipidemia, diabetes, obesity and respiratory conditions, and persons with a diagnosis of cancer or cardiovascular event more than 5 years previously will also be included

Exclusion Criteria:

* new cancer diagnosis or cardiovascular event within 5 years
* alcoholism and alcohol abuse (mild, moderate or severe)
* Unable to participate fully in the program due to mental health or physical limitations
* participating concurrently in other studies of intensive health behaviour modification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in one or more of the Four Core Health Behaviors | 12 weeks, and 3 month follow-up
  Target: at least 150 min moderate to vigorous physical activity and exercise per week .Baseline assumption - 15% of population meets this goal; end of program - at least 30% will meet goal.
  Target: at least 50% reduction in number of smokers
  Reduce long-term health risks by drinking no more than:
  10 drinks a week for women, with no more than 2 drinks a day most days 15 drinks a week for men, with no more than 3 drinks a day most days Target: at least 5 fruits/vegetables per day

SECONDARY OUTCOMES:
Improvement in Risk Factors for Chronic Disease | 12 weeks, and 3 month follow-up
  Blood Pressure: Target <140/90 (<130/80 for persons with DM) Target: at least 10% more people reaching guideline.
  Blood Lipids:Target: at least 10% more people reaching guideline according to their baseline risk category 2nd target: 10% reduction in LDL cholesterol Blood glucose:For persons with diabetes or pre-diabetes, as per CDA guidelines. Target: at least 10% more people reaching guideline for A1C control BMI and Waist Circumference:BMI <25; waist circumference Men: <102 cm Women: <88 cm . Target: at least 10% more people reaching guideline

OTHER OUTCOMES:
Self-efficacy and Behavioural Readiness | 12 weeks, and 3 month follow-up
  Improvement in stage of change by at least one level for key behaviour for that individual

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oh, MD FRCPC, Study Director — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Civljak M, Sheikh A, Stead LF, Car J. Internet-based interventions for smoking cessation. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007078. doi: 10.1002/14651858.CD007078.pub3. PMID 20824856
- [Background] Fraser Health (2013) 'South Asian Health Institute' [Online] Available from: http://www.fraserhealth.ca/about_us/media_centre/news_releases/2013-news-releases/south-asian-health-institute [Accessed March 10, 2013.]
- [Background] Gaikwad R, Warren J. The role of home-based information and communications technology interventions in chronic disease management: a systematic literature review. Health Informatics J. 2009 Jun;15(2):122-46. doi: 10.1177/1460458209102973. PMID 19474225
- [Background] Kisely S, Terashima M, Langille D. A population-based analysis of the health experience of African Nova Scotians. CMAJ. 2008 Sep 23;179(7):653-8. doi: 10.1503/cmaj.071279. PMID 18809896
- [Background] Murray E, Burns J, See TS, Lai R, Nazareth I. Interactive Health Communication Applications for people with chronic disease. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD004274. doi: 10.1002/14651858.CD004274.pub4. PMID 16235356
- [Background] Waters E, de Silva-Sanigorski A, Hall BJ, Brown T, Campbell KJ, Gao Y, Armstrong R, Prosser L, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD001871. doi: 10.1002/14651858.CD001871.pub3. PMID 22161367